CLINICAL TRIAL: NCT01116752
Title: Pediatric ICUs at Emory-Children's Center Glycemic Control: The PedETrol Trial
Brief Title: Pediatric Intensive Care Units (ICUs) at Emory-Children's Center Glycemic Control: The PedETrol Trial
Acronym: PedETrol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB00005792; RO1 (Other: HL096871); Pedetrol5792 (Other: Other)
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Pediatric Patient (1m-21y); ICU Admission; Hyperglycemia
Keywords: Intensive Care; Critical care; Glycemic Control; Hypoglycemia; Hyperglycemia; Insulin treatment; Organ Function; PELOD; Outcomes; Pediatrics
MeSH Terms: conditions — Hyperglycemia; Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strict control (Active Comparator): Children requiring intensive care and mechanical ventilation and/or vasopressor/inotropic support who develop critical illness hyperglycemia (persistent BG values if >140 mg/dL) will be randomized to have their glucose levels managed with insulin infusions and receive strict glycemic control (80-140 mg/dL)
  Interventions: Other: Active Glycemic Control Strict (80-140mg/dL) vs. Conservative (190-220mg/dL) (with or without Continuous Glucose Monitoring)
- Conservative control (Active Comparator): Children requiring intensive care and mechanical ventilation and/or vasopressor/inotropic support who develop critical illness hyperglycemia (persistent BG values if >140 mg/dL) will be randomized to have their glucose levels managed with insulin infusions and receive conservative control (190-220 mg/dL).
  Interventions: Other: Active Glycemic Control Strict (80-140mg/dL) vs. Conservative (190-220mg/dL) (with or without Continuous Glucose Monitoring)

INTERVENTIONS:
Other: Active Glycemic Control Strict (80-140mg/dL) vs. Conservative (190-220mg/dL) (with or without Continuous Glucose Monitoring) — In addition to glycemic control in 2 groups, all children <1 year old and 25% of those >1 year old, will be able to receive continuous glucose monitoring via interstitial glucometry.

SUMMARY:
The primary goal of this project is to determine whether normalizing hyperglycemia is a safe approach to improve multisystem organ function in critically ill children requiring intensive care. The will are conducting the "PedETrol" (the "Pediatric ICUs at Emory-Children's Center Glycemic Control: The PedETrol Trial) Trial, a 4-year single-center, prospective, randomized clinical trial to evaluate the outcome benefit, safety and resource utilization impact of maintaining strict glucose control in children with life-threatening conditions.

***This study is supported by an Research Project Grant (RO1 grant) (MRR) via the National Heart, Lung, and Blood Institute (NHLBI).

DETAILED DESCRIPTION:
Many reports demonstrate improved outcomes in critically ill adults who develop hyperglycemia by rigorous glycemic. Medical oversight committees (including the Institutes of Healthcare Improvement, the American Diabetes Association, and Society of Critical Care Medicine, among others) recommend routine glycemic control during critical illness. Some studies show high rates of hypoglycemia and have highlighted the concern of this approach to care. Little data exists on how hyperglycemia and glycemic control affects critically ill children. Our practice group has developed a regular approach to glycemic control that appears effective and safe and controlling hyperglycemia and the investigators believe that due to our unique experience and expertise in this field, the investigators are well-poised to conduct further much needed studies regarding glycemic control in children. To specifically address the void of knowledge regarding glycemic control in critically ill children, the investigators will conduct a single-center randomized controlled trial to ascertain whether there is vital organ system, outcome, and resource utilization benefit to strict glycemic control vs. more conservative control in children requiring intensive care. The "PedETrol" (the "Pediatric ICUs at Emory-Children's Center Glycemic Control) Trial will study 1,004 children admitted to the ICU for medical, surgical, or cardiac conditions requiring mechanical ventilation and/or vasopressor/i support who develop hyperglycemia, defined as persistent blood glucose >140 mg/dL). Participants will be randomized to either receive strict glycemic control (80-140 mg/dL) or more conservative control (190-220 mg/dL). Insulin infusions will be used to maintain blood glucose in these ranges. In addition to assessing organ and outcome specific efficacy parameters, the investigators will meticulously evaluate for untoward effects including hypoglycemia, and determine the impact of this practice on costly medical resources. All children <1 year old and 25% of those >1 year old, will be able to receive continuous glucose monitoring via interstitial glucometry. This appears to be the first glycemic control trial in any critical care population to make use of continuous glucose monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill children with hyperglycemia, defined as persistent BG >140 mg/dL, meeting the following criteria will be targeted for this study.
* Age 1 month -18 years old
* Admission to the pediatric medical/surgical or pediatric cardiac intensive care unit
* Require mechanical ventilation and/or vasopressors/inotropic infusions
* Patient or family member available to discuss informed consent criteria and provide informed consent.

Exclusion Criteria:

* Age >18 years old
* Age <1 month of chronologic age
* Patients with type I diabetes mellitus or other conditions in which there is impaired glycogen stores or counter regulatory response (i.e. inborn error of metabolism, fulminant hepatic failure)
* Patients with "do not resuscitate", "do not intubate", or "do not escalate care" orders
* Lack of availability by parent or legal guardian to assist in the consent process will be excluded

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 153 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Determine recovery of organ function in critically ill children subject to either strict or conservative glycemic control. | 8/1/2010-3/31/2014
  Determine the rapidity of recovery of organ function in critically ill children subject to either strict or conservative glycemic control by assessing organ function using Pediatric Logistic Organ Dysfunction (PELOD) scoring 6 days following development of hyperglycemia.

SECONDARY OUTCOMES:
Adverse effect rates | 8/1/2010-3/31/2014
  Impact on mortality and other morbidity measures (i.e. ICU length of stay [LOS], mechanical ventilation days, inotrope scores, hospital acquired infections0 1) Adverse effect rates (including moderate (blood glucose [BG] <60 mg/dL) and severe (BG <40 mg/dL) hypoglycemia) associated with strict versus conservative glycemic control in pediatric critical illness.
Glycemic control compared to conservative control on care cost | 8/1/2010-3/31/2014
  Determine the effect of strict glycemic control compared to conservative control on care cost (i.e. hospital and ICU costs) and medical resource utilization (i.e. ICU and mechanical ventilation days) in critically ill children.

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Rigby, MD, PhD, Principal Investigator — Emory University and Children's Healthcare of Atlanta at Egleston
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States

REFERENCES:
- [Background] Preissig CM, Rigby MR, Maher KO. Glycemic control for postoperative pediatric cardiac patients. Pediatr Cardiol. 2009 Nov;30(8):1098-104. doi: 10.1007/s00246-009-9512-4. Epub 2009 Aug 25. PMID 19705188
- [Background] Preissig CM, Rigby MR. Pediatric critical illness hyperglycemia: risk factors associated with development and severity of hyperglycemia in critically ill children. J Pediatr. 2009 Nov;155(5):734-9. doi: 10.1016/j.jpeds.2009.05.007. Epub 2009 Jul 22. PMID 19628220
- [Background] Preissig CM, Rigby MR. A disparity between physician attitudes and practice regarding hyperglycemia in pediatric intensive care units in the United States: a survey on actual practice habits. Crit Care. 2010;14(1):R11. doi: 10.1186/cc8865. Epub 2010 Feb 3. PMID 20128893
- [Background] Vlasselaers D, Milants I, Desmet L, Wouters PJ, Vanhorebeek I, van den Heuvel I, Mesotten D, Casaer MP, Meyfroidt G, Ingels C, Muller J, Van Cromphaut S, Schetz M, Van den Berghe G. Intensive insulin therapy for patients in paediatric intensive care: a prospective, randomised controlled study. Lancet. 2009 Feb 14;373(9663):547-56. doi: 10.1016/S0140-6736(09)60044-1. Epub 2009 Jan 26. PMID 19176240
- [Background] Preissig CM, Hansen I, Roerig PL, Rigby MR. A protocolized approach to identify and manage hyperglycemia in a pediatric critical care unit. Pediatr Crit Care Med. 2008 Nov;9(6):581-8. doi: 10.1097/PCC.0b013e31818d36cb. PMID 18838924